CLINICAL TRIAL: NCT00161148
Title: Probiotics in Patients With Primary Sclerosing Cholangitis and Inflammatory Bowel Disease- a Randomized Placebo-Controlled Cross-Over Trial
Brief Title: Probiotics in Patients With Primary Sclerosing Cholangitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PBPSC
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2007-01-09 (Estimated); Status verified 2007-01

CONDITIONS: Primary Sclerosing Cholangitis
Keywords: PSC; Liver biochemistry; Probiotics; Pruritus
MeSH Terms: conditions — Cholangitis, Sclerosing; Pruritus | interventions — Probiotics

INTERVENTIONS:
Drug: Probiotics

SUMMARY:
PSC is a progressive liver disease without effective medical treatment. There is often co-existent ulcerative colitis. Probiotics (bacterial food supplements) have been shown to benefit patients with ulcerative colitis. In the current protocol potential beneficial effects of probiotics on liver biochemistry and liver related symptoms as pruritus are being assessed in 12 PSC patients in a randomized controlled cross over study (3 months probiotics, 1 one wash-out and 3 months placebo).

DETAILED DESCRIPTION:
I. INTRODUCTION Primary sclerosing cholangitis (PSC) is a progressive cholestatic liver disease characterized by multifocal strictures of intrahepatic and extrahepatic bile ducts, which frequently leads to biliary cirrhosis and liver failure. The aetiology of PSC is unknown but is thought to be (auto)immune-mediated. Nevertheless, in a number of randomized controlled trials a clear benefit of treatment with various immunosuppressive agents, such as D-penicillamine, methotrexate, corticosteroids or nicotine, could not be demonstrated. Although treatment with ursodeoxycholic acid (UDCA) improves serum liver tests and is prescribed on a large scale for PSC patients, this therapeutic modality may have no beneficial effect on the course of the disease.

70 - 90% of patients with PSC have concurrent inflammatory bowel disease (IBD), mostly ulcerative colitis. Conversely, 7% of patients with IBD have PSC. The close association between inflammatory bowel disease and PSC suggests that substances originating from the inflamed gut may damage the liver and biliary tree. Bacterial products may act as toxic proinflammatory agents. N-formyl L-methionine L-leucine L-tyrosine is a peptide produced by enteric flora. When this peptide was introduced into the colon of rats with colitis, it was absorbed, underwent enterohepatic circulation, and appeared undegraded in bile. Histologic changes in the livers of the rats resembled those in PSC.

Probiotics are beneficial bacteria that are used to redress the bacterial composition of the enteric flora which may be altered in disease. Beneficial effects of probiotics have already been described in diseases such as inflammatory bowel disease, pouchitis and non-alcoholic fatty liver disease. Probiotic bacteria have also been shown to counteract inflammatory processes by enhancing the degradation of enteral antigens, reducing the secretion of inflammatory mediators, thereby modifying in a beneficial way the balance between pro- and anti-inflammatory mediators, and stabilizing gut barrier functions. These effects may benefit PSC patients.

Our hypothesis is that administration of probiotics may improve the composition of the enteric flora and subsequently decrease the release of substances that may be toxic and harmful for the liver and biliary tree in PSC patients. Furthermore, immunological alterations induced by treatment with probiotics may have positive effects in PSC.

II. AIM OF THE STUDY Primary aim: assessment of the effects of treatment with probiotics on serum liver tests.

Secondary aim: assessment of the effects of treatment with probiotics on fatigue and pruritus.

III. DESIGN OF THE STUDY Double-blind randomized cross-over pilot study. Eligible patients will be randomized to treatment with probiotics or placebo for a period of 12 weeks. After a wash-out period of 4 weeks, placebo-treated patients will receive verum and vice versa for another period of 12 weeks.

Dosage of concurrent medication for PSC (UDCA, immunosuppressives) will remain the same during the entire study period.

Patients who are being treated with antibiotics during the study period for more than 1 week will be withdrawn from the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PSC based on characteristic findings on cholangiography, or based on the triad: typical histological findings in a liver biopsy, elevated serum alkaline phosphatase and presence of inflammatory bowel disease
* Presence of inflammatory bowel disease
* elevated serum alkaline phosphatase
* age ≥ 18 years
* informed consent

Exclusion Criteria:

* Pregnancy
* use of probiotics within one month before the study
* use of antibiotics within one month before the study
* a history of bacterial cholangitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12
Dates: Start 2005-01; Study Completion 2006-05

PRIMARY OUTCOMES:
Assessment of the effects of treatment with probiotics on serum liver tests

SECONDARY OUTCOMES:
Assessment of the effects of treatment with probiotics on fatigue and pruritus

CONTACTS AND LOCATIONS:
Overall Officials: Karel v Erpecum, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Liu Q, Duan ZP, Ha DK, Bengmark S, Kurtovic J, Riordan SM. Synbiotic modulation of gut flora: effect on minimal hepatic encephalopathy in patients with cirrhosis. Hepatology. 2004 May;39(5):1441-9. doi: 10.1002/hep.20194. PMID 15122774
- [Background] Lindor KD. Ursodiol for primary sclerosing cholangitis. Mayo Primary Sclerosing Cholangitis-Ursodeoxycholic Acid Study Group. N Engl J Med. 1997 Mar 6;336(10):691-5. doi: 10.1056/NEJM199703063361003. PMID 9041099